CLINICAL TRIAL: NCT00484393
Title: Tetracaine (Ametop®) Compared to Placebo for Reducing Pain Associated With Intramuscular Injection of Palivizumab (Synagis®) - A Pilot Study
Brief Title: Tetracaine Compared to Placebo for Reducing Pain With Palivizumab - A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Brandi Newby, Clinical Pharmacy Specialist, Fraser Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2007-041
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Tetracaine; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetracaine (Experimental): Tetracaine 4% gel 1g applied to injection site
  Interventions: Drug: tetracaine 4% gel
- Placebo (Placebo Comparator): Placebo cream (Aquatain) 1g applied to inejction site
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tetracaine 4% gel — tetracaine applied prior to 1 injection
  Other Names: Ametop
  Arms: Tetracaine
Drug: Placebo — placebo applied prior to 1 injection
  Other Names: Aquatain used as placebo to look like tetracaine
  Arms: Placebo

SUMMARY:
This is a small study known as a pilot study. This pilot study is being done to see if a difference in pain from intramuscular palivizumab injection can be detected if tetracaine a topical numbing gel is used compared to no medication (placebo). If a difference is found in this pilot study, then a larger study may be done to confirm that there is a difference in pain experience.

DETAILED DESCRIPTION:
Objective:

1) To determine if tetracaine 4% gel (Ametop ®) reduces the pain of intramuscular palivizumab compared to placebo for pediatric patients between 1 month and 2 years of age.

Rationale:

Premedication with a systemic analgesic has not been shown to be effective in reducing the pain from an acute localized insult. EMLA and tetracaine have been shown to decrease pain associated with immunizations. EMLA requires a 60 minute application, which decreases the usefulness in a busy clinic. Tetracaine has a quicker onset of action and therefore may be more suitable for use in a busy clinic. Efficacy of tetracaine prior to palivizumab has not been reported and therefore it is not known if it can reduce the pain associated with intramuscular palivizumab injection.

Setting:

Respiratory synctial virus (RSV) clinic in the pediatric outpatient ward at Surrey Memorial Hospital.

Procedure:

A notice will be posted in the RSV clinic inviting parents to contact research staff if interested in participating in this study. When a parent contacts staff about the study, a nurse or pharmacist involved in the study will meet with the parent to review eligibility and obtain informed consent.

Once informed consent obtained subject will be randomized by study pharmacist to receive either tetracaine 4% gel (Ametop®) or placebo before administration of the next palivizumab injection (study injection 1); a 4 block randomization design will be used. At the next injection (study injection 2) the subject will receive either tetracaine or placebo, whichever agent they did not receive at study injection 1. The subjects will serve as their own control.

The placebo (Aquatain; Whitehall-Robins, Mississauga, Ontario, Canada) is visually and cosmetically similar to tetracaine 4% gel. One gram of drug or placebo will be dispensed in unit dose 5mL oral syringes, heat sealed to prevent evaporation and stored in a refrigerator for up to one week, after which it will be discarded if unused and redispensed. Tetracaine is commercially available in 1.5g tubes that produce approximately 1g tetracaine.

On the day of immunization and on arrival to the clinic, a clinic nurse who is unaware of the treatment assignment will apply 1g of tetracaine or placebo to the subject's thigh and cover it with a dressing (opcit; Smith and Nephew). They will record the time of the application of the study gel. The clinic nurse will remove the dressing and study gel after 30-45 minutes and record the time of removal. The gel will be wiped from the skin with a paper tissue. A 4-point scale (none, mild, moderate, and severe) will be used to assess local skin reactions after removing study gel. Immediately before the injection the site will be cleaned with an alcohol swab, then the dose (15mg/kg using current weight) of palivizumab will be administered using a ½ - 5/8 inch 23-25 gauge needle. A RSV clinic nurse will inject palivizumab within several minutes of gel removal; clinic nurses will not be aware of the treatment assignment for the subjects.

Study injection 1 and 2 will be video recorded. A mirror will be mounted so the video recorder can capture the subject's reaction both face on and from the mirror image. The videotape will continue until the subject calms down following the injection. The subject can be held by a parent during the injection and provide whatever usual comfort measures they would provide. Following the injection the parent will be asked questions to determine their interpretation of the subject's pain response to the injections and if there any factors that may affect the pain response.

Once both study injections are completed the video will be reviewed and pain assessed for both injections by the same scorer using FLACC pain scale. The scorer will be one pediatric registered nurse who is competent in completing pain analysis for infants. The scorer will be blind as to which dose is tetracaine and which is placebo.

Data Collection:

The data collected will include the FLACC pain scale, parent assessment of patient's pain, factors affecting pain response, as well as identify adverse effects from tetracaine and placebo.

Sample size and statistical Analysis:

The number of subjects with informed consent will determine sample size. Statistical analysis will involve descriptive statistics only.

Ethics:

Confidentiality will always be maintained. No information as to the identify of the child will be placed on the data collection forms. Every child will be assigned a number to facilitate identification by the researchers. Informed consent will be obtained.

Personnel:

A team consisting of nurses, a physician, and a clinical pharmacist from SMH will conduct the study. All personnel are currently involved in the day-to-day management of these children and have the required expertise in carrying out this project.

Timeline:

The study will be submitted for ethical approval by the research ethics board, Fraser Health in April 2007. After approval anticipate patient enrolment to start in November 2007 and complete enrolment by March 2008. A further 4 months will be needed to analyze the data and prepare a manuscript. Expected completion date for the project is July 2008.

Budget:

No additional costs are expected for this study.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 1 month and 2 years of age receiving palivizumab at Surrey Memorial Hospital for 2 consecutive intramuscular injections during the 2007/8 season
* Parents need to complete informed consent.

Exclusion Criteria:

* Allergy/sensitivity to tetracaine, or ester type anaesthetics.
* Infants who present with fever or illness that prevent administration of palivizumab.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandi D Newby, BScPharm, Principal Investigator — Surrey Memorial Hospital
Locations (1):
- Surrey Memorial Hospital, Surrey, British Columbia, Canada

REFERENCES:
- [Background] Young KD. Pediatric procedural pain. Ann Emerg Med. 2005 Feb;45(2):160-71. doi: 10.1016/j.annemergmed.2004.09.019. PMID 15671974
- [Background] Anand KJ, Hickey PR. Pain and its effects in the human neonate and fetus. N Engl J Med. 1987 Nov 19;317(21):1321-9. doi: 10.1056/NEJM198711193172105. No abstract available. PMID 3317037
- [Background] Weisman SJ, Bernstein B, Schechter NL. Consequences of inadequate analgesia during painful procedures in children. Arch Pediatr Adolesc Med. 1998 Feb;152(2):147-9. doi: 10.1001/archpedi.152.2.147. PMID 9491040
- [Background] Jacobson RM, Swan A, Adegbenro A, Ludington SL, Wollan PC, Poland GA; Vaccine Research Group. Making vaccines more acceptable--methods to prevent and minimize pain and other common adverse events associated with vaccines. Vaccine. 2001 Mar 21;19(17-19):2418-27. doi: 10.1016/s0264-410x(00)00466-7. PMID 11257372
- [Background] Meyerhoff AS, Weniger BG, Jacobs RJ. Economic value to parents of reducing the pain and emotional distress of childhood vaccine injections. Pediatr Infect Dis J. 2001 Nov;20(11 Suppl):S57-62. doi: 10.1097/00006454-200111001-00009. PMID 11704725
- [Background] O'Brien L, Taddio A, Ipp M, Goldbach M, Koren G. Topical 4% amethocaine gel reduces the pain of subcutaneous measles-mumps-rubella vaccination. Pediatrics. 2004 Dec;114(6):e720-4. doi: 10.1542/peds.2004-0722. PMID 15574604
- [Background] Halperin BA, Halperin SA, McGrath P, Smith B, Houston T. Use of lidocaine-prilocaine patch to decrease intramuscular injection pain does not adversely affect the antibody response to diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae type b conjugate and hepatitis B vaccines in infants from birth to six months of age. Pediatr Infect Dis J. 2002 May;21(5):399-405. doi: 10.1097/00006454-200205000-00010. PMID 12150176
- [Background] Zempsky WT, Schechter NL. IMpact-RSV Study Group report. Pediatrics. 1999 Oct;104(4 Pt 1):993-4; author reply 995. No abstract available. PMID 10532865
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetracaine Then Placebo: Tetracaine 4% gel 1g applied to injection site prior to next palivizumab injection after enrollment Placebo cream (Aquatain) 1g applied to inejction site prior to subsequent palivizumab injection (1 month after 1st study injection)
- Placebo Then Tetracaine: Placebo cream (Aquatain) 1g applied to inejction site prior to next palivizumab injection after enrollment Tetracaine 4% gel 1g applied to injection site prior to subsequent palivizumab injection (1 month after 1st study injection)
Period: Overall Study
Arm/Group | Tetracaine Then Placebo | Placebo Then Tetracaine
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tetracaine First: Tetracaine 4% gel 1g applied to injection site first, then placebo with subsequent injection
- Placebo First: Placebo cream (Aquatain) 1g applied to inejction site first, then tetracaine with subsequent injection
- Total: Total of all reporting groups
Arm/Group | Tetracaine First | Placebo First | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Customized [Number; unit: participants]
  2-6 months | 4 | 3 | 7
Sex/Gender, Customized [Number; unit: participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Determine if a Difference in Pain Scale Ratings is Detectable Following Intramuscular Palivizumab Injection That Was Pre-treated With Placebo or Tetracaine.
Description: Parent score 1-10 (1 representing no pain and 10 representing extreme pain) FLACC (Face, Legs, Activity, Cry, Consolability) Score 0-10 (at baseline and post injection) (0 representing no pain and 10 representing extreme pain) Change in FLACC score
Time Frame: 2 visits, 1 month apart
Population: Each participant was evaluated for repsonse following tetracaine and following placebo
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tetracaine | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Parent score | 7.3 [5 to 10] | 7.3 [5 to 10]
  FLACC at baseline | 1.7 [0 to 9] | 1.6 [0 to 6]
  FLACC post injection | 8.4 [6 to 10] | 9.3 [8 to 10]
  Change in FLACC | 6.7 [1 to 9] | 7.7 [3 to 10]

ADVERSE EVENTS:
Arm/Group | Tetracaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetracaine (N=7) | Placebo (N=7)
Local skin reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No